CLINICAL TRIAL: NCT03022604
Title: Pharmacokinetic, Hemodynamic and Ergogenic Assessment of a Pre-Workout Dietary Supplement
Brief Title: Assessment of a Pre-Workout Supplement
Acronym: NB6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Nutrabolt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB2014-0795F
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Exercise Ergogenics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- C4/Generation 4 (Experimental): 12 grams of C4/Generation 4 Extreme
  Interventions: Dietary Supplement: C4/Generation 4
- C450X (Active Comparator): 12 grams of C4X (150% of regular dose)
  Interventions: Dietary Supplement: C450X
- Placebo (Placebo Comparator): 12 grams of flavored dextrose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: C4/Generation 4 — 12 grams of C4/Generation 4
  Arms: C4/Generation 4
Dietary Supplement: C450X — 12 grams of C450X
  Arms: C450X
Dietary Supplement: Placebo — 12 grams of flavored dextrose
  Arms: Placebo

SUMMARY:
This study is assessing the effects of a pre-workout dietary supplement.

DETAILED DESCRIPTION:
The purpose of this study is to examine the acute effects of a pre-workout dietary supplement at a standard dose and one that is delivered at 150% of the standard dose on energy metabolism, cardiovascular hemodynamics, blood metabolites and mental focus.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be apparently healthy males and/or females between the ages of 18 and 40
* Participants must have at least 6 months immediate prior history of resistance training including the bench press and leg press/squat

Exclusion Criteria:

* Participants who have a history of treatment for metabolic disease (i.e., diabetes), hypertension, hypotension, thyroid disease, arrhythmias and/or cardiovascular disease
* Participants who currently use any prescription medication
* Participants who are intolerant to caffeine and/or other natural stimulants
* Participants who are pregnant or lactating women
* Participants who have a history of smoking
* Participants who drink excessively (12 drinks per week)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Effects of a Pre-Workout Dietary Supplement on the Stroop Color and Word Test | Seven Days
Effects of a Pre-Workout Dietary Supplement on the Word Recall Test | Seven Days
Effects of a Pre-Workout Dietary Supplement on VAS Readiness to Perform | Seven Days
Effects of a Pre-Workout Dietary Supplement on anaerobic sprint capacity on a bicycle ergometer | Seven Days
Effects of a Pre-Workout Dietary Supplement on bench press power output | Seven Days
Effects of a Pre-Workout Dietary Supplement on leg press power output | Seven Days
Effects of a Pre-Workout Dietary Supplement on total work on the bench press | Seven Days
Effects of a Pre-Workout Dietary Supplement on total work on the leg press | Seven Days

SECONDARY OUTCOMES:
Effects of a Pre-Workout Dietary Supplement on energy expenditure | Seven Days
Effects of a Pre-Workout Dietary Supplement on heart rate | Seven Days
Effects of a Pre-Workout Dietary Supplement on blood pressure | Seven Days
Effects of a Pre-Workout Dietary Supplement on ECG's | Seven Days
Effects of a Pre-Workout Dietary Supplement on blood lab results | Seven Days

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University

IPD SHARING:
Plan to Share IPD: No